CLINICAL TRIAL: NCT01414894
Title: Intensive Management of Pressure and Volume Expansion in Patients With Subarachnoid Hemorrhage
Acronym: IMPROVES
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Miriam Treggiari, Professor, University of Washington
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 37222-A
Record Dates: First submitted 2010-04-05; First posted 2011-08-11 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal Fluids & Normal Blood Pressure (Active Comparator): Patients are treated with conventional fluid replacement (Normovolemia) and maintenance of blood pressure in a normal range (Conventional Blood Pressure).
  Interventions: Other: Fluid manipulation; Other: Blood Pressure Manipulation
- Increased Fluids & Normal Blood Pressure (Active Comparator): Patients are treated with fluids to achieve higher volume expansion (Hypervolemia) and maintenance of blood pressure in a normal range (Conventional Blood Pressure)
  Interventions: Other: Fluid manipulation; Other: Blood Pressure Manipulation
- Normal Fluids & Higher Blood Pressure (Active Comparator): Patients are treated with conventional fluid replacement (Normovolemia) and maintenance of blood pressure in a higher range (Augmented Blood Pressure).
  Interventions: Other: Fluid manipulation; Other: Blood Pressure Manipulation
- Increased Fluids & Higher Blood Pressure (Active Comparator): Patients are treated with fluids to achieve higher volume expansion (Hypervolemia) and maintenance of blood pressure in a higher range (Augmented Blood Pressure).
  Interventions: Other: Fluid manipulation; Other: Blood Pressure Manipulation

INTERVENTIONS:
Other: Fluid manipulation — Patients are treated with conventional fluid replacement (Normovolemia) or increased the fluid replacement (Hypervolemia) for 10 days.
  Other Names: Hypervolemia; Normovolemia
Other: Blood Pressure Manipulation — Patients are treated with maintenance of blood pressure in a normal range (Conventional Blood Pressure) or increased the blood pressure (Augmented Blood Pressure) for 10 days.
  Other Names: Conventional Blood Pressure; Augmented Blood Pressure

SUMMARY:
The purpose of our study is to determine how well Triple-H works and how safe it is. The investigators are hoping to determine the effects of starting the therapy early and to explore if hypervolemia and/or hypertension are beneficial, and what the optimal target ranges are.

DETAILED DESCRIPTION:
Efficacy of Triple-H therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age more than or equal to 18 years
2. Aneurysmal SAH of any clinical grade
3. Head computed tomography demonstrating SAH
4. Cerebral angiography revealing the presence of cerebral aneurysm(s) in a location that explains the SAH
5. Treatment of aneurysm with clipping or coiling must be carried out prior to randomization and within 72 hours of bleeding
6. Signed consent by study participant or applicable legal representative within 72 hours after SAH

Exclusion Criteria:

1. History of traumatic SAH
2. Non-aneurysmal SAH as indicated by no demonstrable aneurysm by cerebral angiography
3. Presence of an unsecured intracranial aneurysm(s) at risk of rupture that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
4. Delayed referral with clipping/coiling greater than 72 hours after the initial bleeding
5. Time of symptom onset cannot be reliably determined
6. Intracranial hypertension (ICP >25 mm Hg) at the time of screening
7. History within the past six months and/or physical findings on admission of decompensated congestive heart failure (NYHA functional class III or IV, or objective class C or D)
8. Acute, evolving or recent myocardial infarction
9. Cardiac arrhythmia or second and third degree atrio-ventricular block causing hemodynamic instability
10. Chronic renal failure requiring dialysis
11. Suspected or confirmed pregnancy
12. Non English speaking
13. A condition that would preclude the performance of the neurobehavioral test battery due to a prior diagnosis of Alzheimer's disease, stroke, degenerative condition, cerebral tumor, or mental retardation
14. Severe terminal disease with life expectancy less than 6 months
15. Refusal of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Our primary endpoint is to determine the feasibility of the pilot study within the ICU setting and collect preliminary estimates for sample size calculations. | 6 months
  1. Estimation of the eligible population once specific study inclusion & exclusion criteria are applied 2. Estimation of enrollment projections, retention, attrition & losses to follow up; 3. Assessment of compliance with protocol instructions; 4. Evaluation of protocol violations; 5. Achievement of pre-determined hemodynamic goals in each study group.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Treggiari, MD, PhH, MPH, Principal Investigator — University of Washington

REFERENCES:
- [Derived] Togashi K, Joffe AM, Sekhar L, Kim L, Lam A, Yanez D, Broeckel-Elrod JA, Moore A, Deem S, Khandelwal N, Souter MJ, Treggiari MM. Randomized pilot trial of intensive management of blood pressure or volume expansion in subarachnoid hemorrhage (IMPROVES). Neurosurgery. 2015 Feb;76(2):125-34; discussion 134-5; quiz 135. doi: 10.1227/NEU.0000000000000592. PMID 25549192